CLINICAL TRIAL: NCT04717817
Title: The PRIMUS Study: Effect of Pre-operative Inspiratory Muscle Training on Post-operative Pulmonary Recovery and Pulmonary Complications After Cardiac Surgery
Brief Title: Inspiratory Muscle Training Prior to Conventional and Minimal Invasive Heart Surgery
Acronym: PRIMUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of time and personnel
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Hasselt University (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001/20200218
Record Dates: First submitted 2021-01-05; First posted 2021-01-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Bypass Graft Surgery; Valve Replacement; Post-Op Complications; Physiotherapy
Keywords: post-operative complications; inspiratory muscle training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: lungfunction assessor, radiologist (thorax X-ray) and physician (hospital ward) are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: experimental (Experimental): Daily inspiratory muscle training (IMT) using an IMT Threshold device (Philips) prior to surgery
  Interventions: Device: Inspiratory muscle training (IMT) using an IMT Threshold device (Philips)
- Group 2: comparator (Active Comparator): Standard physiotherapy prior to surgery
  Interventions: Other: Standard physiotherapy

INTERVENTIONS:
Device: Inspiratory muscle training (IMT) using an IMT Threshold device (Philips) — Inspiratory muscle training on a daily basis prior to surgery during 2-3 weeks
  Arms: Group 1: experimental
Other: Standard physiotherapy — Standard instructions and physiotherapy prior to surgery during 2-3 weeks
  Arms: Group 2: comparator

SUMMARY:
The main objective of this study is to evaluate the effect of pre-operative Inspiratory muscle training (IMT) using an IMT Threshold device (Philips), on early postoperative lung function recovery and on the occurrence of post-operative pulmonary complications (PPC) after major cardiothoracic surgery with and without sternotomy. As frailty can affect postoperative outcome, the relation between frailty, maximal inspiratory pressure (MIP) and post-operative outcome is investigated additionally.

DETAILED DESCRIPTION:
Patients eligible for cardiac surgery are pre-operatively randomized to standard physiotherapy or daily inspiratory muscle training for a period of 2-3 weeks. One therapy session a week is supervised by a physiotherapist in the IMT group. Post-operative physiotherapy is standardized. Pulmonary function and clinical status are evaluated pre-operatively, and during the early post-operative phase, approximately on the 3th and 6th post-operative day, or when necessary. The occurrence of postopercenterative pulmonary complications is determined using a validated scale, the Melbourne group scale, based on clinical status, chest x-ray and blood tests. Frailty is defined based on the Fried criteria. Two Belgian hospitals are involved in this study: the University Hospital Brussels and the Jessa Hospital (Hasselt), the latter mainly focussing on patients referred for minimal invasive heart surgery (minimally invasive-aortic valve replacement (mini-AVR) and Endoscopic - Atraumatic Coronary Artery Bypass (endo-ACAB).

ELIGIBILITY:
Inclusion Criteria:

* Candidates for coronary artery bypass grafting or minimally invasive valve repair/replacement

Exclusion Criteria:

* Not able to perform pre-operative standard pulmonary function tests
* No understanding of Dutch, French or English and/or no ability to understand verbal instructions regarding the inspiratory muscle training
* Patients who participate in another clinical trial
* Patients suffering from neuromuscular disorders, unstable angina, a history of non-traumatic pneumothorax, chronic obstructive pulmonary disease (COPD) in exacerbation
* Patients in need for urgent surgery (within less than 2 weeks)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function (Volumes) | Prior to pre-operative physiotherapy
  Inspiratory capacity (l), Functional residual capacity (l),Residual volume (l), Total lung capacity (l). Baseline. Diagnosis of normal/obstructive/restrictive lungfunction
Pulmonary function (Volumes) | After 2 weeks of pre-operative physiotherapy (before surgery)
  Inspiratory capacity (l), Functional residual capacity (l), Residual volume (l), Total lung capacity (l).Diagnosis of normal/obstructive/restrictive lungfunction and evolution after pre-operative physiotherapy.
Pulmonary function (Volumes) | approximately 6 days after surgery
  Inspiratory capacity (l), Functional residual capacity (l) ,Residual volume (l),Total lung capacity (l). Diagnosis of normal/obstructive/restrictive lungfunction. Evolution after surgery.
Dynamic pulmonary function | Prior to pre-operative physiotherapy
  Vital capacity (l), FVC: forced vital capacity (l), FEV1: forced expiratory volume in 1 second (l). Baseline. Diagnosis of normal/obstructive/restrictive lungfunction.
Dynamic pulmonary function | After 2 weeks of pre-operative physiotherapy (before surgery)
  Vital capacity (l), FVC: forced vital capacity (l), FEV1: forced expiratory volume in 1 second (l). Diagnosis of normal/obstructive/restrictive lungfunction and evolution after pre-operative physiotherapy.
Dynamic pulmonary function | approximately 6 days after surgery
  Vital capacity (l), FVC: forced vital capacity (l), FEV1: forced expiratory volume in 1 second (l).Diagnosis of normal/obstructive/restrictive lungfunction. Evolution after surgery.

SECONDARY OUTCOMES:
post-operative pulmonary complications | early post-operative period (day0 - day7)
  Melbourne Group Scale (MGS), tool for recognition of postoperative pulmonary complications (PPC), based on 1) Temperature >38◦C 2)White blood cell count >11.2 or the use of respiratory antibiotics 3)Physician diagnosis of pneumonia or chest infection 4)Chest X-ray report of atelectasis/pneumonia 5)Production of purulent (yellow/green)sputum differing from preoperative 6)Positive signs on sputum microbiology 7)SpO2<90% on room air 8)Re-admission to or prolonged stay (over36 hours) on the intensive care unit/highdependency unit for respiratory problems. Postoperative pulmonary complications are defined as a score of four or more positive variables. the occurence of PPC is an endpoint in this study.
Hand grip strength | Prior to pre-operative physiotherapy
  Evaluation of hand grip strength using a Martin Vigorimeter
Hand grip strength | 3 days after surgery
  Evaluation of hand grip strength using a Martin Vigorimeter
Hand grip strength | 6 days after surgery
  Evaluation of hand grip strength using a Martin Vigorimeter
Respiratory Muscle Strength Test | Prior the pre-operative physiotherapy
  Maximum inspiratory pressure (MIP)
Respiratory Muscle Strength Test | After 1 week of pre-operative physiotherapy
  Maximum inspiratory pressure (MIP)
Respiratory Muscle Strength Test | After 2 weeks of pre-operative physiotherapy (before surgery)
  Maximum inspiratory pressure (MIP)
Respiratory Muscle Strength Test | 3 days after surgery
  Maximum inspiratory pressure (MIP)
Respiratory Muscle Strength Test | 6 days after surgery
  Maximum inspiratory pressure (MIP)
CRP | Prior the pre-operative physiotherapy
  C-reactive protein, evaluation inflammatory status
CRP | 3 days after surgery
  C-reactive protein, evaluation inflammatory status
CRP | 6 days after surgery
  C-reactive protein, evaluation inflammatory status

OTHER OUTCOMES:
Frailty | basline, Prior the pre-operative physiotherapy
  Frailty measured by the SHARE-FI, SHARE Frailty instrument

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Verdaet, Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No